CLINICAL TRIAL: NCT01232777
Title: Pan-VEGF Blockade for the Treatment of Retinopathy of Prematurity (BLOCK-ROP)
Acronym: BLOCK-ROP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Vision Research Foundation (Other)
Responsible Party: Principal Investigator, Michael T. Trese, M.D., VitreoRetinal Surgeon & Researcher, Vision Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2010-10-26; First posted 2010-11-02 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of Prematurity; Bevacizumab; Avastin; Vascular Endothelial Growth Factor
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bevacizumab (Avastin) 0.75mg/0.03cc (Active Comparator): 1/3 of study participants will be randomized to this treatment in one eye (study eye) and the other eye will receive laser (fellow eye)
  Interventions: Drug: Bevacizumab
- Bevacizumab (Avastin) 0.625mg/0.025cc (Active Comparator): 1/3 of patients will be randomized to this treatment in 1 eye (study eye) and the other eye will receive laser (fellow eye).
  Interventions: Drug: Bevacizumab
- Laser ablation (Active Comparator): 1/3 of study participants will be randomized to this treatment in both eyes (study eye and fellow eye)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — A single dosage of: 0.625mg(0.025cc)or 0.75mg(0.03cc) will be given intravitreally.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to determine whether a single intravitreal (into the gel of the eye) injection of Avastin 0.625mg or 0.75mg is equivalent (non-inferior) to treatment with standard of care laser in infants with Type I pre-threshold retinopathy of prematurity (ROP) diagnosed at 30-36 weeks gestational age.

DETAILED DESCRIPTION:
Retinopathy of Prematurity (ROP) is a leading cause of blindness in children in developed countries around the world, and an increasing cause of blindness in developing countries.

The retina lines the inside of the eye. It functions as "film" within the camera, which is the eye. When an infant is born prematurely, the vascular network necessary to nourish the retina has not fully developed. As a consequence, in some infants abnormal vessels grow instead of the normal ones--a condition known as ROP. The abnormal vessels carry scar tissue along with them, and may lead to retinal detachment and blindness if the eye is not treated.

The multi-center trial of Cryotherapy for Retinopathy of Prematurity (CRYo-ROP) Study demonstrated that ablation of the peripheral avascular retina reduced the risk of poor structural and visual outcome due to retinal distortion or detachment in ROP (1980's). The ablated retina is not functional and is not amendable to regeneration.

Peripheral retinal ablation is not universally effective in fostering regression of ROP. This is particularly true for an aggressive form of ROP (aggressive posterior ROP, or APROP), which typically afflicts profoundly premature and sick neonates. In this subset of infants, progression of ROP to retinal detachments in both eyes and even blindness may occur despite timely and complete peripheral retinal laser ablation.

RATIONALE:

The development of ROP is largely dependant on vascular endothelial growth factor (VEGF). When an infant is born prematurely, the relatively hyperoxic environment that the baby is introduced to shuts down the production of VEGF. Retinal maturation is thus delayed. Subsequently, at a time when intraocular VEGF levels would be declining late in the third trimester of pregnancy, abnormally high levels of VEGF are seen due to large areas of avascular retina and associated tissue hypoxia.

The availability of FDA-approved drugs for anti-VEGF treatment renders it possible to treat such eye off-label. Available drugs include pegaptanib sodium (Macugen) for partial blockage of VEGF-A, or drugs such a ranibizumab (Lucentis) and bevacizumab (Avastin), which cause complete blockage of VEGF-A.

As VEGF is required in the developing retina for normal angiogenesis, and our goal is not to penetrate tissue, but to block the excessive levels of VEGF trapped within the overlying vitreous which is responsible for the abnormal vasculature in ROP.

For purposes of this study, we have chosen bevacizumab (Avastin) which will: a) attain complete blockage (vs. Macugen) of intravitreal VEGF-A, and b)which is limited in its ability to penetrate tissues because it is a full antibody (vs. Lucentis, an antibody fragment specifically designed for better tissue penetration), and is more likely to restore VEGF homeostasis within the developing retina.

ELIGIBILITY:
Inclusion Criteria:

* Inborn babies at participating NICU's who meet inclusion criteria
* Outborn babies transferred to participating NICU's who meet inclusion criteria
* Type 1 pre-threshold ROP
* No prior treatment
* Post menstrual age less than 36 1/7 weeks
* Post menstrual age greater than 30 weeks

Exclusion Criteria:

* Fatal systemic anomaly
* An ocular anomaly of one or both eye affecting the retina or choroid
* An ocular anomaly precluding use of the RetCam (ex., microphthalmia)
* Neonatologist feels inclusion will unduly challenge the infant
* Refusal of initial consent
* Refusal of subsequent evaluation
* Media opacity precluding fundus visualization (ex., cataract)
* Any ocular or periocular infection(s)

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2015-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
To demonstrate non-inferiority of Anti-VEGF treatment to standard-of-care laser | With patient #58, 116 and 174 (within 3 months after each patient being enrolled)
  It is the intent of this clinical study to develop alternative therapy (a single bevacizumab injection) to standard therapy (laser ablation) and to show that bevacizumab is as safe and efficacious as laser.

SECONDARY OUTCOMES:
Decreased laser ablation and improved vascular maturity | With patient #58, 116 & 174 (within 3 months after each patient being enrolled)
  These 2 end-points will be monitored by evidence of persistent disease and presence/absence of progression to retinal detachment. If either or both of these objectives are not met, it is indicative of failure of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Trese, MD, Principal Investigator — Vision Research Foundation
Locations (19):
- United States (18):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jules Stein Eye Institute, UCLA, Los Angeles, California
  - Eye Insitute at Stanford, Palo Alto, California
  - Bascon Palmer Eye Institute, Miami, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Children's Hospital, Dept. of Ophthalmology, Boston, Massachusetts
  - Associated Retinal Consultants/William Beaumont Hospital, Royal Oak, Michigan
  - Insitute of Ophthalmology and Medical Science, New Jersey Medical School, Newark, New Jersey
  - Department of Ophthalmology, Weill Cornell Medical College, New York, New York
  - Abrahamson Pediatric Eye Institute, Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Midwest Retina, Dublin, Ohio
  - University Hospitals Eye Insitute, Rainbow Babies & Children's Hospital, Mayfield Heights, Ohio
  - St. Christopher's Hospital for Children, Drexel Univ. School of Medicine, Philadelphia, Pennsylvania
  - Austin Retina Associates, Austin, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Moran Eye Center, Salt Lake City, Utah
  - Medical College of Wisconsin--Eye Insititute, Milwaukee, Wisconsin
- Ells Retina Centre, Calgary, Alberta, Canada